CLINICAL TRIAL: NCT06747949
Title: A Multicenter, Open-Label, Long-term, Extension Study to Evaluate the Safety and Tolerability of Dazodalibep in Participants With Sjögren's Syndrome (SS)
Brief Title: A Long-term Extension Study of Dazodalibep in Participants With Sjögren's Syndrome (SS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-DAZ-304; 20230050 (Other: Amgen); 2024-517513-32-00 (Other: EU CT Number)
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sjögren's Syndrome
Keywords: Cluster of differentiation 40 (CD40); Dazodalibep; AMG 611
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dazodalibep (Experimental): Participants who completed the 48-week dazodalibep or placebo treatment in trials HZNP-DAZ-301 or HZNP-DAZ-303 will receive assigned dose Dose A of dazodalibep for an additional 132 weeks.
  Interventions: Drug: Dazodalibep

INTERVENTIONS:
Drug: Dazodalibep — Dazodalibep will be given intravenously (IV).
  Other Names: AMG 611

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of dazodalibep.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participant has provided informed consent before initiation of any study specific activities/procedures.
* Must have been eligible to receive and have received IP (dazodalibep or placebo) and completed the study (through Week 48) in one of the phase 3 SS dazodalibep studies (HZNP-DAZ-301, or HZNP-DAZ-303).
* Must be able to receive Dose 1 of this LTE study at the Week 48 Visit (+28 days) for the prior pivotal phase 3 SS dazodalibep studies (HZNP DAZ-301, or HZNP DAZ-303).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Clinically significant active infection at Day 1, in the opinion of the Investigator, including ongoing and chronic infection requiring antibiotics or antiviral medication.
* Planned participation in another clinical study with an IP or procedure during the LTE study. Other investigational procedures and participation in observational research studies while participating in this study are excluded.
* Any condition or change in health status observed or reported during the phase 3 SS studies (HZNP-DAZ-301, or HZNP-DAZ-303) that, in the opinion of the Investigator or the Sponsor, would interfere with evaluation and interpretation of participant safety or alter the risk-benefit associated with IP administration.
* Planned surgeries or hospitalizations that, in the opinion of the Investigator or the Sponsor, would interfere with evaluation and interpretation of participant safety.
* Individuals who plan to receive live (attenuated) vaccine during the LTE study.
* Female participants of childbearing potential unwilling to use protocol-specified method of contraception during treatment and for an additional 12 weeks after the last dose of investigational product.
* Female participants who are pregnant or lactating or planning to become pregnant during the study.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 844 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2029-12-11 (Estimated); Study Completion 2029-12-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 152 weeks
  Includes treatment emergent serious adverse events (TESAEs) and adverse events of special interest (AESIs).

SECONDARY OUTCOMES:
Number of Participants with Anti-drug Antibodies (ADAs) During the Study | Up to 132 weeks
Plasma Concentration of Dazodalibep | Up to 132 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (144):
- United States (30):
  - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - Arizona Arthritis and Rheumatology Associates - Flagstaff - 399 S Malpais Ln, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Associates - Gilbert - 3645 S Rome St, Gilbert, Arizona
  - Arizona Arthritis and Rheumatology Associates - Glendale - 5681 W Beverly Ln, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Associates - Tucson - 2001 W Orange Grove Rd, Tucson, Arizona
  - Samy Metyas MD Inc, Covina, California
  - UCSD Altman Clinical and Translational Research Institute Building, La Jolla, California
  - Tekton Research, LLC - 2121 E Harmony Rd - PPDS, Fort Collins, Colorado
  - Bradenton Research Center Inc, Bradenton, Florida
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - BayCare Medical Group Primary Care and Rheumatology - Tampa, Tampa, Florida
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Kansas City Physician Partners-8350 N Saint Clair Ave, Kansas City, Missouri
  - Arthritis, Rheumatic & Bone Disease Associates - P, Voorhees Township, New Jersey
  - Duke Early Phase Clinical Research Unit - PPDS, Durham, North Carolina
  - Onsite Clinical Solutions, LLC - Salisbury, Salisbury, North Carolina
  - Arthritis & Osteoporosis Center of Southwest Ohio - Miamisburg, Miamisburg, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - STAT Research-600 Aviator Ct, Vandalia, Ohio
  - Murfreesboro Medical Clinic Westlawn, Murfreesboro, Tennessee
  - Accurate Clinical Management-Baytown, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - R & H Clinical Research-777 S Fry Rd, Katy, Texas
  - Houston Rheumatology & Arthritis Specialists - PLLC - PPDS, Katy, Texas
  - Biopharma Informatic - Ridge Road - PPDS, McAllen, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - DM Clinical Research - Migraine and COPD - PPDS, Tomball, Texas
  - Western Washington Medical Group, Bothell - Rheumatology, Bothell, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (12):
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto CER S.A., Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Quilmes, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Privado de Reumatologia - PPDS, San Miguel de Tucumán, Tucumán Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - Aprillus Asistencia e Investigacion - Terrada 89, Buenos Aires
  - Sanatorio Agote - Swiss Medical Group - PPDS, Buenos Aires
  - Sanatorio Allende S.A.-Hipolito Yrigoyen 384, Córdoba
  - Framingham Centro Médico, La Plata
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan
- The Queen Elizabeth Hospital, Woodville South, South Australia, Australia
- UZ Gent, Ghent, Belgium
- Brazil (3):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
- Clinique de Rhumatologie Du Centre Du Quebec, Trois-Rivières, Quebec, Canada
- Chile (3):
  - Centro de Investigacion de Enfermedades Respiratorias e inmunologicas, Viña del Mar, Región de Valparaíso
  - Enroll SpA - Dr. Manuel Barros Borgono - PPDS, Providencia
  - BIOCINETIC Ltda, Santiago
- Croatia (2):
  - Polyclinic Bonifarm, Zagreb, City of Zagreb
  - University Hospital of Split, Split
- France (5):
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - GHRMSA - Hôpital Emile Muller, Mulhouse
  - AP-HP - Hôpital Saint Antoine, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (4):
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Rheumazentrum Prof. Dr. med. Gunther Neeck-Standort Bad Doberan, Bad Doberan, Mecklenburg-Vorpommern
  - Rheumazentrum Greifswald, Greifswald Hansestadt, Mecklenburg-Vorpommern
  - MVZ Rheuma, Hamburg
- Greece (2):
  - University General Hospital of Larissa, Larissa, Larisa
  - Euromedica Kianous Stavros, Thessaloniki
- Hungary (4):
  - Bekes Varmegyei Kozponti Korhaz, Gyula, Bekes County
  - Vasarhelyi Sarkanyfu Kft., Hódmezovásárhely, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen, Hajdú-Bihar
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet - Albert Flórián út 5-7, Budapest
- Israel (2):
  - Meir Medical Center, Kafr Saba, Central District
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
- Italy (5):
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa
  - AUSL di Reggio Emilia - IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
- Japan (13):
  - Chubu Rosai Hospital, Nagoya-shi, Akita
  - Japan Community Health Care Organization (JCHO) Chukyo Hospital, Nagoya-shi, Akita
  - Hospital of the University of Occupational and Environmental Health, Japan, Kita Kyushu-shi, Hukuoka
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku, Ishikawa-ken
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyôto
  - Kyoto University Hospital, Kyoto, Kyôto
  - Kurashiki Medical Clinic, Kurashiki-Shi, Okayama-ken
  - Saitama Medical University Hospital, Iruma-Gun Moroyama-Machi, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - St. Luke's International Hospital, Chuo-Ku, Tokyo
  - Tokyo Medical Center, Meguro-Ku, Tokyo
- Mexico (4):
  - Mediadvance Clinical S.A.P.I. de C.V., Parques de San Felipe, Chihuahua
  - Centro de Investigación en Artritis y Osteoporosis - PPDS, Mexicali, Estado de Baja California
  - Clinstile, S.A. de C.V., Mexico City
  - Unidad de Atención Medica e Investigación en Salud, Mérida
- New Zealand (3):
  - Optimal Clinical Trials Ltd - PPDS, Auckland, North Island
  - Health New Zealand - Te Whatu Ora - Waikato (Waikato Hospital), Hamilton
  - Aotearoa Clinical Trials Trust- Middlemore Hospital, Papatoetoe
- Peru (3):
  - Clinica San Antonio S.A.C, Trujillo, La Libertad
  - Medicentro Biociencias Peru S.R.L., Pueblo Libre, Lima region
  - Instituto de Ginecologia y Reproduccion - PPDS, Santiago de Surco
- Poland (22):
  - Med-Polonia Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Malopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - Zespol Poradni Specjalistycznych REUMED- Wallenroda 2F/4, Lublin, Lublin Voivodeship
  - MICS Centrum Medyczne Warszawa - MICS - PPDS, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - ARS RHEUMATICA Sp. z o.o., Warsaw, Masovian Voivodeship
  - WIM-PIB, Centralny Szpital Kliniczny MON, Warsaw, Masovian Voivodeship
  - Centrum Medyczne K2J2 - Wołomin, Wołomin, Masovian Voivodeship
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. Z o.o., Malbork, Pomeranian Voivodeship
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Katowice - PPDS, Katowice
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow
  - FutureMeds - Lodz - PPDS, Lodz
  - Twoja Przychodnia PCM, Poznan
  - FutureMeds - Warszawa Centrum - PPDS, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu - Borowska 213, Wroclaw
  - Pracownia Badan Klinicznych Salus - ul. Ołtaszyńska 92c/3, Wroclaw
  - FutureMeds - Wroclaw - PPDS, Wroclaw
- Portugal (4):
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon, Lisbon District
  - ULS de Santa Maria,EPE - Hospital de Santa Maria - PPDS, Lisbon, Lisbon District
  - Hospital Conde de Bertiandos - Unidade Local de saúde do Alto Minho, EPE - Ponte de Lima, Ponte de Lima
  - ULS de Gaia/Espinho, EPE - Unidade I, Vila Nova de Gaia
- Serbia (5):
  - Military Medical Academy, Belgrade, Belgrade
  - Institute of Rheumatology - PPDS, Belgrade
  - Klinika za Alergologiju i Imunologiju, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
- University Clinical Centre Maribor, Maribor, Slovenia
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi, South Korea
- Spain (6):
  - Fundacio Hospital de l'Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Universitario de Valme, Seville
- Taiwan (4):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital - PPDS, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (3):
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Chapel Allerton Hospital - PPDS, Leeds
  - Mile End Hospital - PPDS, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code were provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com